CLINICAL TRIAL: NCT00468871
Title: A Multicenter, Randomized, Controlled Study to Evaluate the Safety and Efficacy of an Intravitreal Fluocinolone Acetonide (0.5mg) Implant Compared to Standardized Therapy in Subjects With Non-Infectious Uveitis Affecting the Posterior Segment of the Eye
Brief Title: Safety and Efficacy of Fluocinolone Acetonide Intravitreal Implant vs Standardized Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 415-002
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Non-infectious Uveitis
MeSH Terms: interventions — Fluocinolone Acetonide; Adrenal Cortex Hormones; Immunosuppressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluocinolone acetonide (Experimental): Intravitreal fluocinolone acetonide implant
  Interventions: Drug: fluocinolone acetonide intravitreal implant
- Standard care (Active Comparator): Standard of Care
  Interventions: Drug: corticosteroids and immunosuppressants

INTERVENTIONS:
Drug: fluocinolone acetonide intravitreal implant — surgical intravitreal implant of fluocinolone acetonide
  Arms: Fluocinolone acetonide
Drug: corticosteroids and immunosuppressants — Systemic corticosteroids alone or combined with immunosuppressants
  Arms: Standard care

SUMMARY:
This is a 3 year,superiority, multicenter, open-label, randomised controlled safety and efficacy study. The aim of this study is to evaluate the effect of an intravitreal fluocinolone acetonide (0.59 mg) implant compared to standardized therapy in subjects with unilateral or bilateral, non-infectious uveitis affecting the posterior segment of the eye.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females at least 6 years of age
* History of recurrent unilateral or asymmetric non-infectious posterior uveitis of at east 1 year duration not associated with significant systemic activity of the disease
* The more severely affected eye having had at least 2 separate recurrences
* The more severely affected eye having been treated by systemic therapy for at least one month just before inclusion
* Visual acuity (VA) of at least 1.4 logMAR units at enrollment
* At time of enrollment, </=10 anterior chamber cells/HPF and vitrous haze</= grade 2.

Exclusion Criteria:

* known allergy or contraindication to fluocinolone acetonide, systemic corticosteroids, or the immunosuppressive agents to be administered
* history of retinal detachment, retinoschisis in the area of implantation, or media opacity precluding evaluation of the retina and vitreous
* presence or history of uncontrolled IOP while on steroid therapy resulting in loss of vision, or IOP >25 mm Hg requiring at least 2 types of antiglaucoma medication to be reduced to <25 mm Hg
* history of NIPU only or iritis only with no vitritis, macular edema, vitreous cells, or vitreous haze
* infectious etiology, vitreous hemorrhage, or a toxoplasma scar in the study eye
* ocular surgery and/or trauma on the study eye within 3 months prior to enrollment, or trabeculoplasty or yttrium aluminum garnet laser within 1 month prior to study enrollment
* monocularity
* AIDS
* pregnancy/lactation
* potential for noncompliance
* or participation in other clinical studies within 1 month of enrollment.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2002-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of uveitis in the study eye. | 2 years

SECONDARY OUTCOMES:
The proportion of subjects with a visual acuity improvement of more than 15 letters on ETDRS charts from baseline. | 33 months
Number of recurrences | 33 months
Number of recurrences compared to the 52 weeks prior to enrollment | 33 months
Change in quality of life indices | 33 months
Adjunctive treatment required | 33 months
Change in the size, if present at baseline, of the area of CME on fluorescein angiography | 33 months
Analysis of safety variables | 33 months
Percent of subjects who had at least one recurrence | 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Pavesio, MD, Principal Investigator — Medical Retina Service/Moorfields Eye Hospital

REFERENCES:
- [Background] Jaffe GJ, Martin D, Callanan D, Pearson PA, Levy B, Comstock T; Fluocinolone Acetonide Uveitis Study Group. Fluocinolone acetonide implant (Retisert) for noninfectious posterior uveitis: thirty-four-week results of a multicenter randomized clinical study. Ophthalmology. 2006 Jun;113(6):1020-7. doi: 10.1016/j.ophtha.2006.02.021. Epub 2006 May 9. PMID 16690128
- [Derived] Pavesio C, Zierhut M, Bairi K, Comstock TL, Usner DW; Fluocinolone Acetonide Study Group. Evaluation of an intravitreal fluocinolone acetonide implant versus standard systemic therapy in noninfectious posterior uveitis. Ophthalmology. 2010 Mar;117(3):567-75, 575.e1. doi: 10.1016/j.ophtha.2009.11.027. Epub 2010 Jan 15. PMID 20079922